CLINICAL TRIAL: NCT05836844
Title: APAS Study: Pragmatic Evaluation of the Performance and Safety of the Anchorsure System® Transvaginal Device for Surgical Treatment of Apical Prolapse in Women. A Post-market Multicentre Prospective Observational Cohort Study.
Brief Title: Pragmatic Evaluation of Performance and Safety of the Anchorsure® Transvaginal Device for Surgical Treatment of Apical Prolapse in Women
Acronym: APAS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Lille (Other); Kremlin-Bicetre Hospital, Paris (Unknown); Clinique Sainte-Anne, Strasbourg (Unknown); Centre Hospitalier de La Rochelle (Other)
Responsible Party: Sponsor
Other Study IDs: IDIL/2022/RdT01 2023-A00289-36
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prolapse; Female; Prolapse Uterovaginal; Prolapse; Cervix
Keywords: pelvic organ prolapse
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: The Anchorsure System® — Sacrospinous ligament fixation performed with the Anchorsure Device

SUMMARY:
Pelvic Organ Prolapse affects 50% of parous women, and apical prolapse is one of the most common types of prolapse. Treatment for apical prolapse ranges from observation, non-surgical treatment or surgical repair. An anchoring device can reduce dissection and operative time and is meant to provide strong fixation whilst minimizing potential postoperative pain by avoiding neurovascular injuries. These potential advantages must be evaluated in terms of performance and safety. This cohort study will be on patients undergoing sacrospinous fixation with the Anchorsure® system with a follow-up of 36 months.

DETAILED DESCRIPTION:
Pelvic Organ Prolapse affects 50% of parous women, and apical prolapse is one of the most frequent. Treatment options for women with apical prolapse range from observation, non-surgical treatment or surgical repair. The use of an anchoring device reduces dissection and operative time and is supposed to provide a strong fixation while minimizing potential postoperative pain by avoiding neurovascular injuries. These potential advantages have to be evaluated in terms of performance and safety. This is a cohort study on patients undergoing sacrospinous fixation with the Anchorsure® system with a follow-up of 36 months.The primary objective of the study is to evaluate the performance of the Anchorsure System® for sacrospinous suspension 12 months after surgical treatment of women with apical prolapse in real-life settings.

ELIGIBILITY:
Inclusion Criteria:

* Women with pelvic organ prolapse with leading edge at or beyond the hymen as confirmed by the pelvic organ prolapse quantification system (POP-Q), i.e. Ba ≥ -1 cm for the anterior compartment, and/or Bp ≥ -1 cm for the posterior compartment, and/or C ≥ -1 cm for the apical compartment including recurrence.
* Women due for POP surgery using the Anchorsure System® for apical prolapse suspension with or without concomitant native tissue repair, with or without concomitant hysterectomy and with or without concomitant sling for stress urinary incontinence.
* All women who have not indicated any objection to participating in the study.
* All women who have been correctly informed.

Exclusion Criteria:

* Patient taking part or having taken part in a device or drug interventional study within the last three months (except for VIGI-MESH national registry).
* Patients due for pelvic organ prolapse repair without apical suspension or with anything other than native tissue repair and the Anchorsure System®.
* Patients with uncontrolled diabetes mellitus.
* Patients with active non-controlled or chronic gynaecologic or urinary tract infection and/or local tissue necrosis.
* Patients with ongoing pelvic organ cancer (e.g. uterine, ovarian, bladder, cervix …).
* Patients with a history of radiotherapy in the pelvic area.
* Patients on therapy with immunosuppressive or immunomodulatory treatment within the previous month.
* patients under ongoing oral anticoagulant therapy.
* Patients with stage 0 and 1 pelvic organ prolapse at the time of surgery
* Patients with a preoperative infection contraindicating the surgery

Min Age: 50 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have biological female reproductive organs.
Study Population: The target population is the population of adult women, undergoing a surgical treatment of The target population is the population of adult women, undergoing a surgical treatment for pelvic organ prolapse using Anchorsure System® in the participating centres: Nîmes University Hospital, Lille University Hospital, Sainte-Anne Clinic in Strasbourg, La Rochelle Hospital and Kremlin-Bicêtre Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Successful performance after sacrospinous fixation of the Anchorsure System®. | 12 months after fixation
  YES /NO

SECONDARY OUTCOMES:
Device or procedure-related adverse events: Daily Pain score | Day 0 to Day 30
  All procedure-related adverse events and complications will be recorded using the Clavien-Dindo classification system with a one-month pain diary (filled in once a day using a visual analog scale of 0 to 10 for buttock pain;
Device or procedure-related adverse events: Anchor palpability | 36 months after surgery
  The anchor palpability score will be recorded regularly for up to 36 months after surgery.
Device or procedure-related adverse events: Abnormal findings on clinical examination | 36 months after surgery
  All abnormal findings on clinical examination will be reported including suture exposure, anchor extrusion into another organ, perforation, organ or vascular or nerve injury/damage, fistula, bleeding including hematoma (requiring transfusion or not), thrombotic event, neuromuscular problems (including pain), pelvic discomfort or pain, de novo dyspareunia, infection (e.g. vaginal, urinary tract infection), urinary tract complications including ureteric disorders, urinary retention requiring drainage > 48h, urge symptoms or incontinence (worsening or de novo), de novo constipation or faecal incontinence. Incidences of adverse events will be determined overall, by type of adverse event, severity, compartment and type of sacrospinous suspension (uni versus bilateral and anterior versus posterior).
Type of sacrospinous fixation technique used | Day 0
  The type of sacrospinous fixation technique used: uni/bilateral, anterior/posterior will be recorded
Success of the intervention | 36 months after surgery
  Success is defined as per primary objective and assessed at 36 months after surgery; compartments treated: anterior, apical, posterior, total; type of prolapse: primary or recurrent prolapse.
Complications/adverse events | 36 months after surgery
  Collection of all complications/adverse events up to 36 months after surgery.
Severity of adverse events | 36 months after surgery
  Determination of the level of severity of the adverse event: mild, moderate, severe.
Compartments treated | 36 months after surgery
  Compartments treated: anterior, apical, posterior, total; type of sacrospinous suspension: uni/bilateral, anterior/posterior.
Potential risk factors for the success/failure of the treatment at baseline: Age | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: The patient's age will be recorded
Potential risk factors for the success/failure of the treatment at baseline: Body Mass Index | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: the patient's Body Mass Index will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Previous history of pelvic surgery | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: Any history of pelvic surgery will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Chronic constipation | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: Any history of chronic constipation will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Chronic pulmonary conditions | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: Any history of chronic pulmonary conditions will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Vaginal compartment | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: Details of the patient's vaginal compartment will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Type of prolapse | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: The type of prolapse (recurrent or primary) will be recorded.
Potential risk factors for the success/failure of the treatment at baseline: Pelvic organ Prolapse Q grade | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: the patient's Pelvic Organ Prolapse (POPQ) grade will be recorded as follows :
  Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen Stage 2 the most distal portion of the prolapse is 1 cm or less proximal or distal to the hymenal plane Stage 3 the most distal portion of the prolapse protrudes more than 1 cm below the hymen but protrudes no farther than 2 cm less than the total vaginal length (for example., not all of the vagina has prolapsed) Stage 4 vaginal eversion is essentially complete
Potential risk factors for the success/failure of the treatment at baseline: Concomitant surgery | Day 0
  Collection of potential risk factors for the success/failure of the treatment at baseline: details of any concomitant surgery will be recorded.
Potential risk factors for the occurrence of complications: Age | Day 0
  The patient's age will be recorded in years
Potential risk factors for the occurrence of complications: Body Mass Index | Day 0
  The patient's body mass index (BMI) will be calculated and recorded. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Potential risk factors for the occurrence of complications: Smoking. | Day 0
  The patient's smoking status will be recorded (Regular smoker/Weaned/Number of cigarettes per day/week).
Potential risk factors for the occurrence of complications: Sexual intercourse. | Day 0
  The frequency of the patient's sexual intercourse will be recorded.
Potential risk factors for the occurrence of complications: concomitant surgery | Day 0
  All details of any concomitant surgery in non-target compartment, other concomitant surgery i.e. hysterectomy, mid uretral sling for SUI, etc…will be recorded.
Evolution of the PFDI-20 quality of life score | Day 0
  The Pelvic Floor Distress inventory (PFDI) includes 20 questions. Each question begins with a "yes" or "no" response. If "yes," the patient must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100. The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
Evolution of the PFDI-20 quality of life score | Up to 36 months after surgery.
  The Pelvic Floor Distress inventory (PFDI) includes 20 questions. Each question begins with a "yes" or "no" response. If "yes," the patient must indicate how much bowl, bladder, or pelvic symptoms have been bothering them in the past 3 months on a 4-point scale that ranges from "not at all" (0) to "quite a bit" (4). The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100. The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
Evolution of quality of life scores : PFIQ-7 | Day 0
  The Pelvic Floor Impact Questionnaire-7 (PFIQ-7), a shortened, less comprehensive version of the Pelvic Floor Impact Questionnaire (PFIQ), is a questionnaire about the social impact of the patient's pelvic floor disorders. It consistś of 7 questions and 3 columns, with each question addressing the impact of urinary symptoms, digestive symptoms, and symptoms directly related to prolapse.
Evolution of quality of life scores : PFIQ-7 | Up to 36 months after surgery.
  The Pelvic Floor Impact Questionnaire-7 (PFIQ-7), a shortened, less comprehensive version of the Pelvic Floor Impact Questionnaire (PFIQ), is a questionnaire about the social impact of the patient's pelvic floor disorders. It consistś of 7 questions and 3 columns, with each question addressing the impact of urinary symptoms, digestive symptoms, and symptoms directly related to prolapse.
Evolution of quality of life scores : PISQ-IR | Day 0
  The Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, Revised by the International UroGynocological Association (PISQ-IR) is a disease-specific tool for evaluating the sexual function in women with pelvic floor disorders. It is useful in screening for sexual disorders in women with Urinary Incontinence (UI), pelvic organ prolapse (POP), and anal incontinence. It is used to assess the impact of pelvic floor disorders on female sexual activity and inactivity.
Evolution of quality of life scores : PISQ-IR | Up to 36 months after surgery.
  The Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, Revised by the International UroGynocological Association (PISQ-IR) is a disease-specific tool for evaluating the sexual function in women with pelvic floor disorders. It is useful in screening for sexual disorders in women with Urinary Incontinence (UI), pelvic organ prolapse (POP), and anal incontinence. It is used to assess the impact of pelvic floor disorders on female sexual activity and inactivity.
Patient satisfaction | Up to 36 months after surgery.
  Patient satisfaction will be recorded on a Visual Analog Scale with scores ranging from 0= Extremely Dissatisfied to 6= Extremely Satisfied.
Global impression of improvement (PGI-I) | Up to 36 months after surgery
  The Patient Global impression of improvement (PGI-I) is a scale to describes how the patient's post-operative condition is compared with how it was before surgery:
  Very much better = 1, Much better = 2, A little better = 3, No change = 4, A little worse = 5, Much worse = 6, Very much worse = 7
Frequency of revision and/or surgical re-intervention | Up to 36 months
  The frequency of revision and/or surgical re-intervention including anti-incontinence surgery after sacrospinous suspension will be recorded

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - La Rochelle General Hospital, La Rochelle
  - Lille University Hospital, Lille
  - Kremlin-Bicêtre Hospital, Paris
  - Clinique Sainte-Anne, Strasbourg